CLINICAL TRIAL: NCT03302026
Title: A Proof-of-concept Study of Real-time fMRI Neurofeedback Training for Smoking Cessation
Brief Title: Real Time fMRI and Quitting Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 828012
Record Dates: First submitted 2017-09-26; First posted 2017-10-04 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Nicotine Use Disorder
Keywords: nicotine treatment; real time fMRI
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: The proposed study will evaluate the effects of rt-fMRI neurofeedback training on the ability to resist craving for cigarettes. The study will be conducted in two phases: a technical development phase and a proof-of-concept phase focused on efficacy. The technical development phase will be completed before beginning the proof-of-concept phase. Eligible consenting treatment-seeking smokers complete an intake session and then be randomized to an active NFT group or a control group. Both groups will complete three scanning sessions, followed by a smoking resist evaluation.
Who Masked: Participant
Masking Description: Treatment-seeking smokers complete an intake session and then be randomized to an active NFT group or a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-time neurofeedback training group (Experimental): We propose to use rt-fMRI neurofeedback training to help smokers consciously modulate activation in areas related to cravings and self-control in order to improve control smoking urges. In this arm, participants will complete four sessions: an intake session and 3 neurofeedback scanning visits. The primary outcome is the ability to resist smoking during a validated smoking lapse paradigm. Secondary outcomes include changes in brain activity in areas related to craving and self-control, and self-reported craving for cigarettes.
  Interventions: Behavioral: Realtime biofeedback using fMRI
- No-feedback control group (No Intervention): We propose to use rt-fMRI neurofeedback training to help smokers consciously modulate activation in areas related to cravings and self-control in order to improve control smoking urges. In the control group arm, participants will complete four sessions: an intake session and 3 scanning visits with no neurofeeback. The primary outcome is the ability to resist smoking during a validated smoking lapse paradigm. Secondary outcomes include changes in brain activity in areas related to craving and self-control, and self-reported craving for cigarettes.

INTERVENTIONS:
Behavioral: Realtime biofeedback using fMRI — Real-time fMRI (rt-fMRI) allows for rapid analysis of brain activation while an individual is actively performing a task, and can be used to provide real-time neurofeedback to individuals during fMRI scanning. Using neurofeedback, individuals can learn to modulate activity in specific regions of the brain. We propose to use rt-fMRI neurofeedback training to help smokers consciously modulate activation in areas related to cravings and self-control in order to improve control smoking urges. Participants will complete four sessions: an intake session and 3 scanning visits. The primary outcome is the ability to resist smoking during a validated smoking lapse paradigm.
  Arms: Real-time neurofeedback training group

SUMMARY:
This study will examine how real-time functional magnetic resonance imaging (rt-fMRI) feedback can be used to modulate brain activation in the context of smoking cues in order to resist craving. Participants will complete a total of three fMRI scanning sessions with a cue suppression task with or without neurofeedback training (NFT). Participants will be randomized to an active group (active NFT) or a control group (no NFT) during the scanning sessions. At the end of the third session, all participants will complete a validated smoking lapse laboratory paradigm to evaluate effects of NFT on smoking behavior.

DETAILED DESCRIPTION:
Smoking is the greatest preventable cause of mortality and a significant economic burden. Even with the best available treatments, most smokers relapse within days or weeks after a quit attempt. Nicotine replacement therapy, the most widely used pharmacotherapy, yields end of treatment quit rates of <25% suggesting that managing nicotine withdrawal is not sufficient. A smoker's response to smoking cues is one factor that increases risk of relapse. This study will examine how real-time functional magnetic resonance imaging (rt-fMRI) feedback can be used to modulate brain activation in the context of smoking cues in order to resist craving. First, we will conduct a pilot study in 12 smokers for technical development and to evaluate the feasibility of the proposed study procedures. Participants will complete a total of three fMRI scanning sessions with a cue suppression task with or without neurofeedback training (NFT). Participants will be randomized to an active group (active NFT) or a control group (no NFT) during the scanning sessions. At the end of the third session, all participants will complete a validated smoking lapse laboratory paradigm to evaluate effects of NFT on smoking behavior. Upon successful completion of the technical development phase, we will proceed to a proof-of-concept phase, which will recruit 72 smokers to evaluate the efficacy of NFT for smoking behavior.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment-seeking smokers between the ages of 18 and 65, reporting consumption of at least 10 cigarettes per day for at least the past 6 months;
2. Planning to live in the area for at least the next month;
3. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form;
4. Able to communicate fluently in English (speaking, writing, and reading).

Exclusion Criteria:

Smoking Behavior:

1. Use of chewing tobacco or snuff or cigars;
2. Current enrollment or plans to enroll in another smoking cessation program or research study in the next month;
3. Current or anticipated (within the next month) use of smoking cessation medications or nicotine replacement therapy (NRT);
4. A baseline carbon monoxide (CO) reading less than 10ppm.

Alcohol/Drugs:

1. Current alcohol consumption that exceeds 25 standard drinks/week;
2. Positive breath alcohol concentration test (BrAC greater than or equal to 0.01) at intake; a. Participants testing positive for breath alcohol with a reading equal to or greater than .08 (the legal driving limit) or who are visibly impaired will be instructed not to drive themselves home after the appointment. If a participant needs to use a phone to call for a safe ride home, an office telephone will be made available to the participant.

Medication:

Current use or recent discontinuation (within the past 30 days at the time of Intake) of:

1. Smoking cessation medication (e.g., Zyban, Wellbutrin, Wellbutrin SR, Chantix, NRT);
2. Anti-psychotic medications;
3. Any medication that could compromise participant safety as determined by the Principal Investigator and/or Study Physician;

   Daily use of:
4. Opiate-containing medications for chronic pain.

Medical/Neuropsychiatric:

1. Women who are pregnant, planning a pregnancy, and/or breast feeding. All female subjects of childbearing potential will undergo a urine pregnancy test at Intake and at each scan session.
2. History of epilepsy or a seizure disorder;
3. History of stroke;
4. Self-reported brain (or CNS) or spinal tumor;
5. Self-reported history of head trauma;
6. Self-reported history or current diagnosis of psychosis.

fMRI-Related:

1. Self-reported use of pacemakers, certain metallic implants, or presence of metal in the eye as contraindicated for fMRI;
2. Self-reported history of claustrophobia;
3. Being left-handed;
4. Color blindness;
5. Weight greater than 250lbs at intake;
6. Self-reported history of gunshot wounds;
7. Any impairment preventing participants from using the response pad necessary for the computer tasks;
8. Circumstances or conditions that may interfere with magnetic resonance imaging (MRI).

General Exclusion:

1. Any medical condition, illness, disorder, or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator;
2. Enrollment or plans to enroll in another research study;
3. Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Smoking Lapse Paradigm | Study session 3 (scan day 3)
  Time (sec) to first cigarette during a 50 minute monitored smoking lapse period in smoking laboratory

SECONDARY OUTCOMES:
Cue induced brain signal change | Study session 3 (scan day 3)
  Change in mean percent signal change for Cue minus Neutral contrasts in activated brain regions

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided